CLINICAL TRIAL: NCT05137496
Title: A Single-center, Prospective, Non-comparative Clinical Trial of Ruxolitinib and Methylprednisolone as a First-line Treatment for Macrophage Activation Syndrome
Brief Title: Ruxolitinib and Methylprednisolone as a First-line Treatment for Macrophage Activation Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Clinical Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ruxolitinib-steroids-MAS
Record Dates: First submitted 2021-11-24; First posted 2021-11-30 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Macrophage Activation Syndrome
MeSH Terms: conditions — Macrophage Activation Syndrome | interventions — ruxolitinib; Methylprednisolone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib+methylprednisolone (Experimental): Ruxolitinib and methylprednisolone administered as the first-line therapy
  Interventions: Drug: Ruxolitinib; Drug: methylprednisolone

INTERVENTIONS:
Drug: Ruxolitinib — 0.3mg/kg/d, iv.gtt, for at least 2 weeks
Drug: methylprednisolone — 2mg/kg, d1-d5, gradually reduced, for at least 2 weeks

SUMMARY:
The present study was a single-center, prospective, non-comparative in which macrophage activation syndrome patients were selected as the main subjects to evaluate the effect and safety of Ruxolitinib and methylprednisolone regimens as the first-line therapy .

ELIGIBILITY:
Inclusion Criteria:

1. Meet hemophagocytic lymphohistiocytosis (HLH)-04 diagnostic criteria; patients were diagnosed with autoimmune disease associated HLH (Macrophage activation syndrome, MAS).
2. No HLH induction therapy was performed.
3. The expected survival time is more than 1 month.
4. Serum creatinine ≤ 1.5 times normal；Serum human immunodeficiency virus(HIV) antigen or antibody negative； Hepatitis C virus (HCV) antibody is negative, or HCV antibody is positive, but HCV RNA is negative；HBV copies less than 1E+03 copies/ml.
5. Total bilirubin ≤10 times the upper limit of normal; serum creatinine ≤1.5 times the normal value
6. The left ventricular ejection fraction (LVEF) was normal.
7. No uncontrollable infection.
8. Contraception for both male or female.
9. Informed consent obtained.

Exclusion Criteria:

1. Pregnancy or lactating Women；
2. Allergic to ruxolitinib；
3. Active bleeding of the internal organs；
4. uncontrollable infection；
5. Serious mental illness;
6. Non-melanoma skin cancer history;
7. Patients unable to comply during the trial and/or follow-up phase;
8. Participate in other clinical research at the same time.

Ages: 1 Year to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Response rate | Change from before and 2,4,6 and 8 weeks after initiating Ruxolitinib combined with methylprednisolone therapy
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.
Progression Free Survival | 2 years
  from date of inclusion to date of progression, relapse, or death from any cause
Adverse events | 2 years
  Adverse events including myelosuppression, infection, hemorrhage

IPD SHARING:
Plan to Share IPD: Undecided